CLINICAL TRIAL: NCT02253992
Title: A Phase 1/2 Dose Escalation and Cohort Expansion Study of the Safety and Tolerability of Urelumab Administered in Combination With Nivolumab in Advanced/Metastatic Solid Tumors and B-cell Non-Hodgkins Lymphoma
Brief Title: An Investigational Immuno-therapy Study to Determine the Safety of Urelumab Given in Combination With Nivolumab in Solid Tumors and B-cell Non-Hodgkin's Lymphoma
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CA186-107; 2014-002241-22 (EudraCT Number)
Record Dates: First submitted 2014-09-29; First posted 2014-10-01 (Estimated); Results first posted 2020-10-05 (Actual); Last update posted 2020-10-05 (Actual); Status verified 2020-09

CONDITIONS: Advanced Solid Tumors; Advanced B-cell NHL
MeSH Terms: interventions — urelumab; Nivolumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Dose Escalation and Cohort expansion: Urelumab + Nivolumab (Experimental): Nivolumab followed by Urelumab
  Nivolumab every 2 weeks up to 12 cycles and Urelumab every 4 weeks up to 6 cycles
  Interventions: Biological: Urelumab; Biological: Nivolumab

INTERVENTIONS:
Biological: Urelumab
  Other Names: BMS-663513
Biological: Nivolumab
  Other Names: BMS-936558

SUMMARY:
The purpose of this study is to determine which doses of Urelumab and Nivolumab are safe and tolerable when they are given together.

ELIGIBILITY:
For more information regarding BMS clinical trial participation, please visit www.BMSStudyConnect.com

Inclusion Criteria:

* For Dose Escalation:

  * Subjects with any previously treated advanced (metastatic or refractory) solid tumor type and B-cell non-Hodgkin lymphoma
* For Cohort Expansion:

  * Subjects must have a previously treated advanced solid tumor or B cell non-Hodgkin's lymphoma to be eligible
  * Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
  * For certain subjects, willing and able to provide pre-treatment and on-treatment fresh tumor biopsy
  * Women of child-bearing potential and men must use an acceptable method of contraception during treatment and for 23 weeks after treatment for women and 31 weeks for men

Exclusion Criteria:

* Known central nervous system metastases or central nervous system as the only source of disease
* Other concomitant malignancies (with some exceptions per protocol)
* Active, known or suspected autoimmune disease
* Uncontrolled or significant cardiovascular disease
* History of hepatitis (B or C)
* History of active or latent tuberculosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 232 (Actual)
Dates: Start 2014-09-29 (Actual); Primary Completion 2019-05-24 (Actual); Study Completion 2019-05-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (17):
- United States (11):
  - Stanford University School Of Medicine, Palo Alto, California
  - H. Lee Moffitt Cancer Center, Tampa, Florida
  - University Of Chicago, Chicago, Illinois
  - Johns Hopkins Sidney Kimmel Comprehensive Cancer Center, Lutherville, Maryland
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - NYU Langone Medical Center, New York, New York
  - Memorial Sloan Kettering Nassau, New York, New York
  - Providence Portland Medical Center, Portland, Oregon
  - UPMC Cancer Center, Pittsburgh, Pennsylvania
  - Md Anderson, Houston, Texas
- France (4):
  - Local Institution, Besançon
  - Local Institution, Marseille
  - Local Institution, Rennes
  - Local Institution, Villejuif
- Universitaetsklinikum Essen, Essen, Germany
- Clinica Universidad de Navarra, Pamplona, Spain

REFERENCES:
- [Derived] Khushalani NI, Ott PA, Ferris RL, Cascone T, Schadendorf D, Le DT, Sharma MR, Barlesi F, Sharfman W, Luke JJ, Melero I, Lathers D, Neely J, Suryawanshi S, Sanyal A, Holloway JL, Suryawanshi R, Ely S, Segal NH. Final results of urelumab, an anti-CD137 agonist monoclonal antibody, in combination with cetuximab or nivolumab in patients with advanced solid tumors. J Immunother Cancer. 2024 Mar 7;12(3):e007364. doi: 10.1136/jitc-2023-007364. PMID 38458639
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.bmsstudyconnect.com/s/US/English/USenHome
- See also: Investigator Inquiry Form — https://www.bms.com/researchers-and-partners/investigator-inquiry-form.html
- See also: FDA Safety Alerts and Recalls — https://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 160 enrolled and treated
Groups:
- TRT A: URE3 Q4WK+NIV3 Q2WK
- TRT B: URE8 Q4WK+NIV3 Q2WK
- TRT D: URE8 Q4WK+NIV240mg Q2WK
Period: Overall Study
Arm/Group | TRT A | TRT B | TRT D
Started | 6 | 4 | 150
Completed (Completed= Continuing in the treatment period.) | 0 | 0 | 6
Not Completed | 6 | 4 | 144
Not completed — Study drug toxicity | 1 | 0 | 10
Not completed — Disease progression | 4 | 3 | 98
Not completed — Withdrawal by Subject | 0 | 0 | 3
Not completed — Adverse Event | 0 | 0 | 8
Not completed — Death | 0 | 0 | 1
Not completed — Subject discontinued study drug | 1 | 0 | 1
Not completed — Completed treatment as per protocol | 0 | 1 | 22
Not completed — Other | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: All treated participants
Groups:
- Total: Total of all reporting groups
Arm/Group | TRT A | TRT B | TRT D | Total
Number analyzed (Participants) | 6 | 4 | 150 | 160
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 1 | 2 | 67 | 70
  >=65 years | 5 | 2 | 83 | 90
Age, Continuous [Mean (Standard Deviation); unit: Years] | 64.7 (9.40) | 64.0 (8.52) | 63.8 (11.71) | 63.9 (11.52)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 47 | 51
  Male | 4 | 2 | 103 | 109
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1 | 2
  Not Hispanic or Latino | 5 | 2 | 107 | 114
  Unknown or Not Reported | 1 | 1 | 42 | 44
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 9 | 9
  White | 6 | 4 | 136 | 146
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 4 | 4

OUTCOME MEASURES:

1. Primary Outcome: The Incidence of Adverse Events.
Time Frame: From day 1 until 100 days after participant last dose of study drug.
Population: All treated participants
Measure: Number; unit: Number of participants
Arm/Group | TRT A | TRT B | TRT D
Number analyzed (Participants) | 6 | 4 | 150
Number of participants | 6 | 4 | 150

2. Primary Outcome: The Incidence of Seriuos Adverse Events.
Time Frame: From day 1 until 100 days after participant last dose of the study drug.
Population: All treated participants
Measure: Number; unit: Number of participants
Arm/Group | TRT A | TRT B | TRT D
Number analyzed (Participants) | 6 | 4 | 150
Number of participants | 3 | 3 | 86

3. Primary Outcome: The Incidence of Death.
Time Frame: From day 1 until 100 days after participant last dose of study drug.
Population: All Treated participants
Measure: Number; unit: Number of participants
Arm/Group | TRT A | TRT B | TRT D
Number analyzed (Participants) | 6 | 4 | 150
Number of participants | 6 | 2 | 93

4. Secondary Outcome: Best Overall Response (BOR)
Description: The total number of subjects whose best overall response (BOR) is either a complete response or partial response for solid tumors and complete remission or partial remission for B-cell NHL, divided by the total number of subjects in the population of interest.
Time Frame: Every 8 weeks for Cycle 1 through Cycle 6 then every 12 weeks thereafter for approximately 2 years.
Population: All treated Participants
Measure: Number; unit: Number of participants
Groups:
- TRT D - NSCLC pd1/Pd-l1 Experienced: URE8 Q4WK+NIV240mg Q2WK- Non small cell lung cancer pd1/pd-l1 experienced
- TRT D - NSCLC pd1/Pd-l1 Naive: URE8 Q4WK+NIV240mg Q2WK - Non samll cell lung cancer pd1/pd-l1 naive.
- TRT D - Melanoma pd1/Pd-l1 Experienced: URE8 Q4WK+NIV240mg Q2WK - Melanoma pd1/pd-l1 experienced
- TRT A - Melanoma pd1/Pd-l1 Naive: URE3 Q4WK+NIV3 Q2WK - Melanoma pd1/pd-l1 naive
- TRT B -: URE8 Q4WK+NIV3 Q2WK - Melanoma pd1/pd-l1 naive
- TRT D - Melanoma pd1/Pd-l1 Naive: URE8 Q4WK+NIV240mg Q2WK - Melanoma pd1/pd-l1 naive
- TRT A - SCCHN: URE3 Q4WK+NIV3 Q2WK - Squamous cell carcinoma of head and neck.
- TRT D - SCCHN: URE8 Q4WK+NIV240mg Q2WK - Squamous cell carcinoma of head and neck.
- TRT A - Other Solid Tumors: URE3 Q4WK+NIV3 Q2WK - Other solid tumors
- TRT B - Other Solid Tumors: URE8 Q4WK+NIV3 Q2WK - Other Solid tumors.
- TRT D - DLBCL: URE8 Q4WK+NIV240mg Q2WK - Diffuse Large B-cell lymphoma.
- TRT D - FL: URE8 Q4WK+NIV240mg Q2WK - Follicular Lymphoma.
Arm/Group | TRT D - NSCLC pd1/Pd-l1 Experienced | TRT D - NSCLC pd1/Pd-l1 Naive | TRT D - Melanoma pd1/Pd-l1 Experienced | TRT A - Melanoma pd1/Pd-l1 Naive | TRT B - | TRT D - Melanoma pd1/Pd-l1 Naive | TRT A - SCCHN | TRT D - SCCHN | TRT A - Other Solid Tumors | TRT B - Other Solid Tumors | TRT D - DLBCL | TRT D - FL
Number analyzed (Participants) | 20 | 20 | 20 | 4 | 1 | 43 | 1 | 21 | 1 | 3 | 22 | 4
Number of participants
  Complete response | 0 | 0 | 0 | 0 | 1 | 6 | 0 | 1 | 0 | 0 | 0 | 0
  Partial response | 1 | 1 | 2 | 1 | 0 | 15 | 0 | 0 | 0 | 0 | 0 | 0

5. Secondary Outcome: Objective Response Rate (ORR)
Description: Objective response rate (ORR) is defined as the total number of subjects whose BOR is either CR or PR divided by the total number of subjects in the population of interest.
Time Frame: Every 8 weeks for Cycle 1 through Cycle 6 then every 12 weeks thereafter for approximately 2 years.
Population: All treated Participants
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | TRT D - NSCLC pd1/Pd-l1 Experienced | TRT D - NSCLC pd1/Pd-l1 Naive | TRT D - Melanoma pd1/Pd-l1 Experienced | TRT A - Melanoma pd1/Pd-l1 Naive | TRT B - | TRT D - Melanoma pd1/Pd-l1 Naive | TRT A - SCCHN | TRT D - SCCHN | TRT A - Other Solid Tumors | TRT B - Other Solid Tumors | TRT D - DLBCL | TRT D - FL
Number analyzed (Participants) | 20 | 20 | 20 | 4 | 1 | 43 | 1 | 21 | 1 | 3 | 22 | 4
Percentage of participants | 5.0 [0.1 to 24.9] | 5.0 [0.1 to 24.9] | 10.0 [1.2 to 31.7] | 25.0 [0.6 to 80.6] | 100.0 [2.5 to 100.0] | 48.8 [33.3 to 64.5] | 0 [0.0 to 97.5] | 4.8 [0.1 to 23.8] | 0 [0.0 to 97.5] | 0 [0.0 to 70.8] | 0 [0.0 to 16.1] | 0 [0.0 to 60.2]

6. Secondary Outcome: Occurrence of Specific Anti-drug Antibodies (ADA) to Urelumab and Nivolumab
Time Frame: Cycles 1, 2, 3, 4, 6, and followup Days up to 100 days.
Population: All treated participants
Measure: Number; unit: Number of participants
Groups:
- Urelumab ADA: Urelumab Anti drug antibody
- Nivolumab ADA: Nivolumab anti drug antibody
Arm/Group | Urelumab ADA | Nivolumab ADA
Number analyzed (Participants) | 133 | 128
Number of participants
  Baseline ADA positive | 5 | 2
  ADA positive | 55 | 9
  ADA negative | 78 | 119

7. Secondary Outcome: Duration of Response (DOR)
Description: DOR is defined as the number of days between the date of first response and the subsequent date of objectively documented disease progression based on the criteria (RECIST v1.1) or relapse based on IWG, or death due to any cause, if death occurred within 100 days after last dose, whichever occurs first.
  Data was not collected due to discontinuation of the study/Due to study termination.
Time Frame: Every 8 weeks for Cycle 1 through Cycle 6 then every 12 weeks thereafter for approximately 2 years
Population: Data was not collected due to discontinuation of the study/Due to study termination.
Arm/Group | TRT A | TRT B | TRT D
Number analyzed (Participants) | 0 | 0 | 0

8. Secondary Outcome: Progression-free Survival Rate (PFSR)
Description: PFSR is defined as the probability of a subject remaining progression-free and surviving a specific length of time.
  Data was not collected due to discontinuation of the study/Due to study termination.
Time Frame: Every 8 weeks for Cycle 1 through Cycle 6 then every 12 weeks thereafter for approximately 2 years.
Population: Data was not collected due to discontinuation of the study/Due to study termination.
Arm/Group | TRT A | TRT B | TRT D
Number analyzed (Participants) | 0 | 0 | 0

9. Secondary Outcome: Maximum Observed Serum Concentration (Cmax)
Description: Data was not collected due to discontinuation of the study/Due to study termination.
Time Frame: Cycles 1, 2, 3, 4, 6, and followup Days up to 100 days.
Population: Data was not collected due to discontinuation of the study/Due to study termination.
Arm/Group | TRT A | TRT B | TRT D
Number analyzed (Participants) | 0 | 0 | 0

10. Secondary Outcome: Time of Maximum Observed Serum Concentration (Tmax)
Description: Data was not collected due to discontinuation of the study/Due to study termination.
Time Frame: Cycles 1, 2, 3, 4, 6, and followup Days up to 100 days.
Population: Data was not collected due to discontinuation of the study/Due to study termination.
Arm/Group | TRT A | TRT B | TRT D
Number analyzed (Participants) | 0 | 0 | 0

11. Secondary Outcome: Area Under the Concentration-time Curve in One Dosing Interval (AUCTAU)
Description: Data was not collected due to discontinuation of the study/Due to study termination.
Time Frame: Cycles 1, 2, 3, 4, 6, and followup Days up to 100 days
Population: Data was not collected due to discontinuation of the study/Due to study termination.
Arm/Group | TRT A | TRT B | TRT D
Number analyzed (Participants) | 0 | 0 | 0

12. Secondary Outcome: Trough Observed Plasma Concentration(Ctrough)
Description: Data was not collected due to discontinuation of the study/Due to study termination.
Time Frame: Cycles 1, 2, 3, 4, 6, and followup Days up to 100 days.
Population: Data was not collected due to discontinuation of the study/Due to study termination.
Arm/Group | TRT A | TRT B | TRT D
Number analyzed (Participants) | 0 | 0 | 0

13. Secondary Outcome: End of Infusion Concentration (Ceoinf)
Description: Data was not collected due to discontinuation of the study/Due to study termination.
Time Frame: Cycles 1, 2, 3, 4, 6, and followup Days up to 100 days.
Population: Data was not collected due to discontinuation of the study/Due to study termination.
Arm/Group | TRT A | TRT B | TRT D
Number analyzed (Participants) | 0 | 0 | 0

14. Secondary Outcome: Area Under the Plasma Concentration-time Curve, 0 to Time of Last Quantifiable Concentration (AUC(0-T)
Description: Data was not collected due to discontinuation of the study/Due to study termination.
Time Frame: Cycles 1, 2, 3, 4, 6, and followup Days up to 100 days.
Population: Data was not collected due to discontinuation of the study/Due to study termination.
Arm/Group | TRT A | TRT B | TRT D
Number analyzed (Participants) | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: From the start dosing day and up to 100 days after participant's last dose ( up to 3 years).
Arm/Group | TRT A | TRT B | TRT D
All-Cause Mortality (participants affected / at risk) | 6/6 | 2/4 | 93/150
Serious Adverse Events (participants affected / at risk) | 3/6 | 3/4 | 86/150
Other Adverse Events (participants affected / at risk) | 6/6 | 4/4 | 147/150
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | TRT A (N=6) | TRT B (N=4) | TRT D (N=150)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 2
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 1
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 2
Atrial flutter (Cardiac disorders) | 0 | 0 | 1
Atrioventricular block (Cardiac disorders) | 0 | 0 | 1
Stress cardiomyopathy (Cardiac disorders) | 0 | 0 | 1
Diabetes insipidus (Endocrine disorders) | 0 | 0 | 1
Hypogonadism (Endocrine disorders) | 0 | 0 | 1
Hypophysitis (Endocrine disorders) | 0 | 0 | 1
Hypothyroidism (Endocrine disorders) | 0 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 3
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 2
Colitis (Gastrointestinal disorders) | 1 | 0 | 1
Constipation (Gastrointestinal disorders) | 0 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 1
Diverticulum intestinal haemorrhagic (Gastrointestinal disorders) | 0 | 0 | 1
Enteritis (Gastrointestinal disorders) | 1 | 0 | 0
Faecaloma (Gastrointestinal disorders) | 0 | 0 | 1
Ileus (Gastrointestinal disorders) | 1 | 0 | 0
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 0 | 3
Asthenia (General disorders) | 0 | 0 | 1
Fatigue (General disorders) | 0 | 0 | 1
General physical health deterioration (General disorders) | 1 | 0 | 4
Hyperthermia (General disorders) | 0 | 0 | 1
Hypothermia (General disorders) | 0 | 0 | 1
Pain (General disorders) | 0 | 0 | 4
Pelvic mass (General disorders) | 0 | 0 | 1
Pyrexia (General disorders) | 0 | 0 | 5
Sudden death (General disorders) | 0 | 0 | 1
Autoimmune hepatitis (Hepatobiliary disorders) | 0 | 0 | 1
Bile duct stenosis (Hepatobiliary disorders) | 1 | 0 | 0
Contrast media reaction (Immune system disorders) | 0 | 0 | 1
Drug hypersensitivity (Immune system disorders) | 0 | 0 | 1
Haemophagocytic lymphohistiocytosis (Immune system disorders) | 0 | 0 | 1
Bacteraemia (Infections and infestations) | 0 | 0 | 1
Bronchitis (Infections and infestations) | 0 | 0 | 1
Cellulitis (Infections and infestations) | 0 | 0 | 1
Device related infection (Infections and infestations) | 0 | 0 | 1
Erysipelas (Infections and infestations) | 0 | 0 | 1
Lung infection (Infections and infestations) | 0 | 0 | 3
Pneumonia (Infections and infestations) | 0 | 0 | 4
Pneumonia haemophilus (Infections and infestations) | 0 | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 0 | 1
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Tracheal obstruction (Injury, poisoning and procedural complications) | 0 | 0 | 1
Alanine aminotransferase increased (Investigations) | 0 | 0 | 2
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 2
Blood alkaline phosphatase increased (Investigations) | 0 | 0 | 1
Blood bilirubin increased (Investigations) | 0 | 0 | 1
Gamma-glutamyltransferase increased (Investigations) | 0 | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 1 | 0 | 1
Diabetes mellitus (Metabolism and nutrition disorders) | 0 | 0 | 1
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 0 | 0 | 1
Failure to thrive (Metabolism and nutrition disorders) | 0 | 0 | 3
Gout (Metabolism and nutrition disorders) | 0 | 0 | 1
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Abdominal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 2
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 37
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Metastases to lymph nodes (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 3
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 3
Ataxia (Nervous system disorders) | 0 | 0 | 1
Central nervous system lesion (Nervous system disorders) | 0 | 1 | 0
Cerebral haematoma (Nervous system disorders) | 0 | 0 | 1
Cerebrovascular accident (Nervous system disorders) | 0 | 0 | 1
Dizziness (Nervous system disorders) | 0 | 0 | 1
Monoplegia (Nervous system disorders) | 0 | 0 | 1
Paraparesis (Nervous system disorders) | 0 | 0 | 1
Seizure (Nervous system disorders) | 0 | 0 | 3
Syncope (Nervous system disorders) | 0 | 0 | 3
Confusional state (Psychiatric disorders) | 0 | 1 | 1
Mental status changes (Psychiatric disorders) | 0 | 0 | 1
Persistent depressive disorder (Psychiatric disorders) | 0 | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 1 | 0 | 1
Haematuria (Renal and urinary disorders) | 0 | 0 | 1
Hydronephrosis (Renal and urinary disorders) | 1 | 0 | 0
Urinary tract obstruction (Renal and urinary disorders) | 0 | 0 | 1
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Hydrothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2
Obstructive airways disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Pharyngeal haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 4
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 3
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 3
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Embolism (Vascular disorders) | 0 | 0 | 1
Extremity necrosis (Vascular disorders) | 0 | 0 | 1
Peripheral ischaemia (Vascular disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | TRT A (N=6) | TRT B (N=4) | TRT D (N=150)
Anaemia (Blood and lymphatic system disorders) | 3 | 1 | 47
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 8
Adrenal insufficiency (Endocrine disorders) | 1 | 0 | 2
Hypothyroidism (Endocrine disorders) | 0 | 1 | 16
Dry eye (Eye disorders) | 0 | 1 | 5
Lacrimation increased (Eye disorders) | 0 | 1 | 2
Vision blurred (Eye disorders) | 2 | 0 | 2
Abdominal discomfort (Gastrointestinal disorders) | 0 | 1 | 0
Abdominal distension (Gastrointestinal disorders) | 1 | 0 | 6
Abdominal pain (Gastrointestinal disorders) | 2 | 1 | 19
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0 | 6
Anal incontinence (Gastrointestinal disorders) | 1 | 0 | 1
Ascites (Gastrointestinal disorders) | 0 | 1 | 0
Constipation (Gastrointestinal disorders) | 1 | 0 | 31
Dental caries (Gastrointestinal disorders) | 0 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 5 | 0 | 32
Dry mouth (Gastrointestinal disorders) | 1 | 0 | 8
Dysphagia (Gastrointestinal disorders) | 2 | 1 | 6
Gastritis (Gastrointestinal disorders) | 1 | 0 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 1 | 3
Lip swelling (Gastrointestinal disorders) | 0 | 1 | 0
Melaena (Gastrointestinal disorders) | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 3 | 0 | 37
Vomiting (Gastrointestinal disorders) | 3 | 0 | 26
Asthenia (General disorders) | 1 | 1 | 16
Chills (General disorders) | 0 | 0 | 14
Fatigue (General disorders) | 4 | 2 | 61
Gait disturbance (General disorders) | 1 | 0 | 1
Oedema peripheral (General disorders) | 1 | 0 | 25
Performance status decreased (General disorders) | 0 | 1 | 1
Pyrexia (General disorders) | 4 | 1 | 29
Hepatic haemorrhage (Hepatobiliary disorders) | 1 | 0 | 0
Gastroenteritis (Infections and infestations) | 1 | 0 | 0
Gingivitis (Infections and infestations) | 1 | 0 | 1
Localised infection (Infections and infestations) | 1 | 0 | 0
Nasopharyngitis (Infections and infestations) | 0 | 1 | 6
Pneumonia (Infections and infestations) | 1 | 0 | 4
Upper respiratory tract infection (Infections and infestations) | 1 | 0 | 12
Urinary tract infection (Infections and infestations) | 1 | 0 | 12
Fall (Injury, poisoning and procedural complications) | 1 | 1 | 8
Infusion related reaction (Injury, poisoning and procedural complications) | 0 | 1 | 2
Skin abrasion (Injury, poisoning and procedural complications) | 0 | 1 | 1
Sunburn (Injury, poisoning and procedural complications) | 0 | 1 | 1
Alanine aminotransferase increased (Investigations) | 2 | 0 | 26
Amylase increased (Investigations) | 0 | 0 | 13
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 26
Blood alkaline phosphatase increased (Investigations) | 2 | 0 | 20
Blood creatinine increased (Investigations) | 1 | 0 | 8
Blood thyroid stimulating hormone increased (Investigations) | 0 | 1 | 4
Blood uric acid decreased (Investigations) | 1 | 0 | 1
Gamma-glutamyltransferase increased (Investigations) | 2 | 0 | 18
Lipase increased (Investigations) | 1 | 0 | 17
Lymphocyte count decreased (Investigations) | 2 | 0 | 7
Neutrophil count decreased (Investigations) | 1 | 0 | 3
Platelet count decreased (Investigations) | 1 | 0 | 8
Weight decreased (Investigations) | 1 | 0 | 18
Decreased appetite (Metabolism and nutrition disorders) | 2 | 1 | 24
Dehydration (Metabolism and nutrition disorders) | 1 | 0 | 4
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 8
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 14
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 0 | 11
Hypermagnesaemia (Metabolism and nutrition disorders) | 1 | 0 | 1
Hyperuricaemia (Metabolism and nutrition disorders) | 1 | 0 | 2
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 0 | 12
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 1 | 9
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 | 0 | 4
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 14
Hypophosphataemia (Metabolism and nutrition disorders) | 2 | 0 | 16
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 2 | 17
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 23
Flank pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 2 | 1 | 5
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 11
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 15
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 6
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 15
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1
Balance disorder (Nervous system disorders) | 0 | 1 | 1
Carotid artery occlusion (Nervous system disorders) | 0 | 1 | 0
Cognitive disorder (Nervous system disorders) | 0 | 1 | 1
Dizziness (Nervous system disorders) | 1 | 0 | 13
Headache (Nervous system disorders) | 4 | 0 | 23
Peripheral motor neuropathy (Nervous system disorders) | 1 | 0 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 1 | 0 | 3
Restless legs syndrome (Nervous system disorders) | 0 | 1 | 1
Sciatica (Nervous system disorders) | 0 | 1 | 0
Sinus headache (Nervous system disorders) | 1 | 0 | 1
Anxiety (Psychiatric disorders) | 0 | 0 | 11
Depression (Psychiatric disorders) | 1 | 0 | 3
Insomnia (Psychiatric disorders) | 0 | 0 | 11
Dysuria (Renal and urinary disorders) | 1 | 0 | 3
Pollakiuria (Renal and urinary disorders) | 1 | 0 | 6
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 33
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 26
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 6
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Actinic keratosis (Skin and subcutaneous tissue disorders) | 1 | 1 | 5
Drug eruption (Skin and subcutaneous tissue disorders) | 1 | 0 | 2
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 13
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Lichen planus (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 2 | 22
Rash (Skin and subcutaneous tissue disorders) | 0 | 1 | 16
Rash macular (Skin and subcutaneous tissue disorders) | 1 | 0 | 2
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 2 | 9
Rash papular (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Rash pruritic (Skin and subcutaneous tissue disorders) | 1 | 0 | 2
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 | 0 | 1
Hot flush (Vascular disorders) | 1 | 0 | 1
Hypertension (Vascular disorders) | 2 | 0 | 3
Hypotension (Vascular disorders) | 1 | 0 | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Statistical Analysis Plan (2016-07-18): https://cdn.clinicaltrials.gov/large-docs/92/NCT02253992/SAP_000.pdf
  • Study Protocol (2017-03-22): https://cdn.clinicaltrials.gov/large-docs/92/NCT02253992/Prot_001.pdf